CLINICAL TRIAL: NCT03001219
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Phase II Study to Evaluate The Safety and Efficacy of RO7123520 as Adjunct Treatment in Patients With Moderately to Severely Active Rheumatoid Arthritis and an Inadequate Response to TNF-alpha Inhibitors
Brief Title: A Study of RO7123520 to Evaluate the Safety and Efficacy in Participants With Moderately To Severely Active Rheumatoid Arthritis (RA) Who Are Inadequately Responding to Anti-Tumor Necrosis Factor (TNF)-Alpha Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was prematurely terminated due to a lack of efficacy of the investigational drug.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP39261; 2016-002126-36 (EudraCT Number)
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Part 1: Placebo (Placebo Comparator): Participants will receive placebo (matched to RO7123520) on Days 1, 14, 28, and 56 with pre-trial anti-TNF-alpha and methotrexate.
  Interventions: Drug: Anti-TNF-alpha; Drug: Methotrexate; Drug: Placebo
- Part 1: RO7123520 (Experimental): Participants will receive RO7123520 on Days 1, 14, 28, and 56 with pre-trial anti-TNF-alpha and methotrexate.
  Interventions: Drug: Anti-TNF-alpha; Drug: Methotrexate; Drug: RO7123520
- Part 2: Placebo (Placebo Comparator): Participants will receive placebo (matched to RO7123520) on Days 1, 14, 28, and 56 with pre-trial anti-TNF-alpha and methotrexate.
  Interventions: Drug: Anti-TNF-alpha; Drug: Methotrexate; Drug: Placebo
- Part 2: RO7123520 (Experimental): Participants will receive RO7123520 on Days 1, 14, 28, and 56 with pre-trial anti-TNF-alpha and methotrexate.
  Interventions: Drug: Anti-TNF-alpha; Drug: Methotrexate; Drug: RO7123520
- Part 3: Placebo (Placebo Comparator): Participants will receive placebo (matched to RO7123520) on Days 1, 14, 28, and 56 with pre-trial anti-TNF-alpha and methotrexate.
  NOTE: Part 3 was not conducted.
  Interventions: Drug: Anti-TNF-alpha; Drug: Methotrexate; Drug: Placebo
- Part 3: RO7123520 (Experimental): Participants will receive RO7123520 on Days 1, 14, 28, and 56 with pre-trial anti-TNF-alpha and methotrexate.
  NOTE: Part 3 was not conducted.
  Interventions: Drug: Anti-TNF-alpha; Drug: Methotrexate; Drug: RO7123520

INTERVENTIONS:
Drug: Anti-TNF-alpha — Participants will continue their pre-trial anti-TNF-alpha therapy at a stable dose.
Drug: Methotrexate — Participants will continue their pre-trial methotrexate therapy at a stable dose.
Drug: Placebo — Participants will receive intravenous infusion of placebo.
  Arms: Part 1: Placebo; Part 2: Placebo; Part 3: Placebo
Drug: RO7123520 — Participants will receive intravenous infusion of RO7123520.
  Arms: Part 1: RO7123520; Part 2: RO7123520; Part 3: RO7123520

SUMMARY:
This is a Phase IIa/b double-blind, placebo-controlled, randomized, parallel group, multicenter study to evaluate the safety and efficacy of RO7123520 as adjunctive therapy in participants with RA who are inadequately responding to standard-of-care (methotrexate and anti-TNF-alpha therapy). Part 1 of the study will evaluate safety. Part 2 will evaluate efficacy and safety. Part 3 will evaluate dose-ranging efficacy. Participants will have the option of continuing to the extension period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult-onset RA as defined by the ACR 2010 criteria, for at least 6 months before screening
* Moderately to severely active RA as defined by at least 4/28 tender joints and at least 4/28 swollen joints, and a DAS28 greater than or equal to (≥) 3.2
* For Part 2 only: Active synovitis and/or osteitis as determined by contrast-enhanced magnetic resonance imaging
* Participants must be taking stable dose of anti-TNF-alpha therapies
* Participants on stable oral glucocorticoids within 6 weeks of planned randomization
* Participants taking non-steroidal anti-inflammatory drugs (NSAIDs) intermittently (up to 2-3 times weekly) for short-term relief of pain and participants on regular NSAID use (on stable dose for ≥ 4 weeks)

Exclusion Criteria:

* Parenteral glucocorticoids administration (intramuscular, IV) of ≥50 mg within 6 weeks or less than or equal to (≤) 50 milligrams (mg) within 4 weeks prior to planned randomization, or scheduled parenteral administrations during the study
* Joint(s) injected with intra-articular glucocorticoids or hyaluronic acid within 6 weeks prior to planned randomization
* Active inflammatory diseases of the joints not related to RA
* Systemic autoimmune disease other than RA
* Juvenile idiopathic arthritis or juvenile RA and/or RA developed before the age of 16
* Active fibromyalgia that makes appropriate assessment of RA disease activity challenging in the opinion of the Investigator
* RA participants functional status class IV according to the ACR 1991 criteria
* Participants with severe chronic or recurrent viral, bacterial, parasitic, or fungal infections
* History of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection
* Any identified confirmed congenital or acquired immunodeficiency
* Abnormal laboratory values and liver function test
* Myocardial infarction within less than 6 months prior to participation in the study
* Severe central or peripheral nervous system diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (80):
- United States (31):
  - Pinnacle Research Group; Llc, Central, Anniston, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Arizona Arthritis and Rheuma, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Medvin Clinical Research, Covina, California
  - University of California San Diego, La Jolla, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Stanford hospital & Clinics; Investigational Drug Services, Stanford, California
  - Omega Research Consultants LLC, DeBary, Florida
  - San Marcus Research Clinic, Inc., Hialeah, Florida
  - Millenium Research, Ormond Beach, Florida
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Shores Rheumatology PC, Saint Clair Shores, Michigan
  - Arthritis & Osteoporosis Associates, Freehold, New Jersey
  - Atlantic Coast Rheumatology, Toms River, New Jersey
  - Ocean Rheumatology, Toms River, New Jersey
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Saint Lawrence Health System; Rheumatology, Canton, New York
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Advanced Rheumatology & Arthritis Research Center, Wexford, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Columbia Arthritis Center (Partnership Practice), Columbia, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Adriana Pop-Moody MD Clinic PA, Corpus Christi, Texas
  - Metroplex Clinical Research, Dallas, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Southwest Rheumatology, Mesquite, Texas
  - Accurate Clinical Research, Inc, Stafford, Texas
- Argentina (4):
  - Centro de Investigaciones Reumatologicas y Osteologicas, Buenos Aires
  - Organización medica de Investi, Cap Fed
  - Cer San Juan, San Juan
  - Centro Medico Privado de Reumatologia; Reumathology, San Miguel
- Medizinische Universität Wien, Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Colombia (6):
  - Centro Integral de Reumatologia del Caribe SAS CIRCARIBE SAS, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialdades Medicas SAS. CIREEM, Bogotá
  - Riesgo de Fractura S.A., Bogotá
  - Fundación Instituto de Reumatología Fernando Chalem, Bogotá
  - Servimed S.A.S., Bucaramanga
  - Healthy Medical Center SAS, Zipaquirá
- Charité Research Organisation GmbH, Berlin, Germany
- Guatemala (2):
  - Centro de Estudio y Tratamiento de Enfermedades Reumaticas, Guatemala City
  - Clinica Privada de Reumatologia Dr. Henry Briones Alvarado, Guatemala City
- Italy (4):
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino; Radiology, Torino, Abruzzo
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola Malpighi; U.O. Malattie Infettive, Bologna, Emilia-Romagna
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliero Universitaria Careggi - SOD Reumatologia, Florence, Tuscany
- Mexico (10):
  - Investigacion y Biomedicina de Chihuahua, Sociedad Civil, Chichuahua, Chihuahua
  - Centro de Investigacion del Noroeste SC, Tijuana, Estado de Baja California
  - Centro Integral en Reumatología S.A. de C.V. (CIRSA), Guadalajara, Jalisco
  - Unidad de Atencion Medica e Investigacion en Salud (UNAMIS), Mérida, Yucatán
  - Centro Médico de las Américas, Mérida, Yucatán
  - Javier Orozco Private Practice, Guadalajara
  - Centro de Investigación; Artritis y Osteoporosis S.C., Mexicali
  - Hospital Angeles Lindavista, México
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - Policlinica Medica de Queretaro S.C., Querétaro
- Peru (4):
  - Hogar Clínica San Juan de Dios, Arequipa
  - Clinica Internacional Sede Lima, Lima
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Instituto de Ginecología y Reproducción, Lima
- Spain (8):
  - Hospital Universitario Marques de Valdecilla; Servicio de Reumatologia, Santander, Cantabria
  - Complexo Hospitalario Universitario A Coruña; Servicio de Reumatología, A Coruña, LA Coruña
  - Hospital de Basurto; Servicio de Reumatologia, Bilbao, Vizcaya
  - Hospital Universitario de la Princesa; Servicio de Reumatologia, Madrid
  - Hospital General Universitario Gregorio Marañon; Servicio de Reumatología, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Psiquiatria, Málaga
  - Hospital Universitario Reina Sofía; Servicio de Aparato Digestivo, Murcia
- United Kingdom (9):
  - New Queen Elizabeth Hospital Birmingham, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - Barts Hospital; Department of Rheumatology, London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Newcastle U. Medical School; Institute of Cellular Medicine, Newcastle
  - University of Oxford, Botnar Research Centre, Oxford
  - Derriford Hospital, Plymouth
  - Lister Hospital; Rheumatology Dept, Stevenage

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult men and women with moderate to severe active rheumatoid arthritis (RA) who experience an inadequate response to disease-modifying anti-rheumatic drug (DMARD) therapy with MTX plus anti-TNF-a therapy.
Pre-assignment Details: Arms are not mutually exclusive.
  Proof of Concept: 109 total participants enrolled.
  Extension Period Analysis: 106 participants from the previous groups, including placebo, received 360 (n=9) or 810 mg/dose (n=97) of RO7123520.
  Part 3 was not conducted due to early study termination.
Groups:
- PoC Placebo to Extension Period Analysis RO7123520: In the Proof of Concept (PoC) period, participants received placebo (IV saline matched to RO7123520) + pre-trial anti-TNF-alpha and methotrexate (MTX), on Days 1, 14, 28, and 56. Participants from this group that continued to the Extension Period Analysis period were assigned RO7123520 + pre-trial anti-TNF-alpha and MTX at either 360 or 810 mg/dose up to Week 20 of the Extension Period (overall study Week 32).
- RO70123520 360 or 810 mg/Dose: In the PoC period, participants not assigned placebo received RO7123520 + pre-trial anti-TNF-alpha and MTX at 810 mg/dose on Days 1, 14, 28, and 56. Participants continuing to the Extension Period Analysis period received 360 or 810 mg/dose up to Week 20 of the Extension Period (overall study Week 32).
Period: Proof of Concept
Arm/Group | PoC Placebo to Extension Period Analysis RO7123520 | RO70123520 360 or 810 mg/Dose
Started | 37 | 72
Completed | 35 | 65
Not Completed | 2 | 7
Not completed — Study Termination by Sponsor | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Protocol Deviation | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 0
Period: Extension Period Analysis
Arm/Group | PoC Placebo to Extension Period Analysis RO7123520 | RO70123520 360 or 810 mg/Dose
Started | 9 | 97
Completed | 4 | 52
Not Completed | 5 | 45
Not completed — Study Termination by Sponsor | 0 | 36
Not completed — Participant Non-Compliance | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Deviation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Population: Proof of Concept: A total of 109 participants were enrolled, 37 in the placebo group and 72 in the 810 mg/dose group.
  Extension Period Analysis: A total of 106 participants from the previous groups received either 360 or 810 mg/dose of RO7123520, with 9 in the 360 mg/dose group and 97 in the 810 mg/dose group.
Groups:
- Total: Total of all reporting groups
Arm/Group | PoC Placebo to Extension Period Analysis RO7123520 | RO70123520 360 or 810 mg/Dose | Total
Number analyzed (Participants) | 37 | 97 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] — Proof of Concept participants Population: The proof of concept groups included 37 participants receiving placebo treatment and 72 participants receiving 810 mg/dose of RO7123520.
  Years
    number analyzed (Participants) | 37 | 72 | 109
    (all) | 54.7 (14.1) | 52.3 (12.3) | 53.1 (13.0)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Extension Period Analysis participants Population: The extension period analysis population contained participants from period 1 of the study. Participants were assigned either 360 (n=9) or 810 (n=97) mg/dose and grouped accordingly.
  Years
    number analyzed (Participants) | 9 | 97 | 106
    (all) | 56.6 (14.3) | 53.4 (12.8) | 53.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Proof of Concept participants Population: The proof of concept groups included 37 participants receiving placebo treatment and 72 participants receiving 810 mg/dose of RO7123520.
  Participants
    number analyzed (Participants) | 37 | 72 | 109
    Female | 32 | 66 | 98
    Male | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants] — Extension Period Analysis participants Population: The extension period analysis population contained participants from period 1 of the study. Participants were assigned either 360 (n=9) or 810 (n=97) mg/dose and grouped accordingly.
  Participants
    number analyzed (Participants) | 9 | 97 | 106
    Female | 6 | 87 | 93
    Male | 3 | 10 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Proof of Concept participants Population: The proof of concept groups included 37 participants receiving placebo treatment and 72 participants receiving 810 mg/dose of RO7123520.
  Participants
    number analyzed (Participants) | 37 | 72 | 109
    Hispanic or Latino | 27 | 54 | 81
    Not Hispanic or Latino | 10 | 18 | 28
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Extension Period Analysis participants Population: The extension period analysis population contained participants from period 1 of the study. Participants were assigned either 360 (n=9) or 810 (n=97) mg/dose and grouped accordingly.
  Participants
    number analyzed (Participants) | 9 | 97 | 106
    Hispanic or Latino | 1 | 73 | 74
    Not Hispanic or Latino | 8 | 24 | 32
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Proof of Concept participants Population: The proof of concept groups included 37 participants receiving placebo treatment and 72 participants receiving 810 mg/dose of RO7123520.
  Participants
    number analyzed (Participants) | 37 | 72 | 109
    American Indian or Alaska Native | 7 | 12 | 19
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 1 | 2
    White | 25 | 52 | 77
    More than one race | 2 | 4 | 6
    Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The extension period analysis population contained participants from period 1 of the study. Participants were assigned either 360 (n=9) or 810 (n=97) mg/dose and grouped accordingly.
  Participants
    number analyzed (Participants) | 9 | 97 | 106
    American Indian or Alaska Native | 0 | 16 | 16
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 7 | 68 | 75
    More than one race | 0 | 6 | 6
    Unknown or Not Reported | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline to last participant last visit (approximately 2 years)
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: In the Proof of Concept (PoC) period, participants received placebo (IV saline matched to RO7123520) + pre-trial anti-TNF-alpha and methotrexate (MTX), on Days 1, 14, 28, and 56.
- Proof of Concept: RO7123520 810mg/Dose: In the PoC period, participants not assigned placebo received RO7123520 + pre-trial anti-TNF-alpha and MTX at 810 mg/dose on Days 1, 14, 28, and 56.
- Extension Period Analysis: RO7123520 360mg/Dose: Participants received 360 mg/dose of RO7123520 + pre-trial anti-TNF-alpha and MTX up to Week 20 of the Extension Period (overall study Week 32).
- Extension Period Analysis: RO70123520 810mg/Dose: Participants received RO7123520 + pre-trial anti-TNF-alpha and MTX at 810 mg/dose up to Week 20 of the Extension Period (overall study Week 32).
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 70 | 9 | 97
Percentage of Participants | 48.6 | 60.0 | 66.7 | 60.8

2. Primary Outcome: Proportion of Participants Achieving an American College of Rheumatology (ACR) 50 Response at Week 12
Description: The ACR50 is a composite measure defined as both improvement of 50% in the number of tender and number of swollen joints, and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP). The ACR is reported as percent improvement at discrete time points.
Time Frame: Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants. Overall study = up to 32 weeks per participant. PoC = Weeks 1-12, Extension Period Analysis = Weeks 1-20 (overall study weeks 13-32)
Measure: Number (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 72 | 9 | 97
Percent | 16.2 [7.67 to 29.95] | 11.1 [5.86 to 19.48] | 0 [0 to 30.89] | 1.0 [0.07 to 5.28]

3. Primary Outcome: Percentage of Participants With Anti-Drug Antibodies
Time Frame: Baseline
Population: This outcome measure only includes the immunogenicity population, which was the PoC 810 mg dose group. These participants had at least 1 pre-dose ADA assessment.
Measure: Number; unit: Percent
Arm/Group | Proof of Concept: RO7123520 810mg/Dose
Number analyzed (Participants) | 69
Percent | 0

4. Primary Outcome: Change From Baseline in Bone Mineral Density Lumbar Spine L1-L4 as Assessed by Dual Energy X-ray Absorptiometry (DEXA) Scans
Time Frame: Baseline, Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 70 | 9 | 97
g/cm^2
  Baseline: number analyzed (Participants) | 37 | 67 | 9 | 94
  Baseline | 1.02 (0.21) | 2.51 (12.46) | 1.17 (0.20) | 2.06 (10.53)
  Week 12: number analyzed (Participants) | 32 | 59 | 6 | 72
  Week 12 | -0.06 (0.20) | 0.71 (5.50) | -0.01 (0.04) | 0.58 (4.98)

5. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Week 12
Description: The CDAI for Rheumatoid Arthritis (RA) assesses the severity of the disease using clinical data. It consists of the Patient Global disease Activity (PGA) estimate and the Evaluator Global disease Activity (EGA) estimate, each of which represent assessments of disease activity on a scale of 1-10, with 10 being maximum activity.
Time Frame: Baseline, Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 72 | 9 | 97
Units on a scale
  Baseline: number analyzed (Participants) | 37 | 69 | 9 | 96
  Baseline | 37.05 (10.99) | 37.38 (13.14) | 30.89 (15.31) | 32.17 (15.91)
  Week 12: number analyzed (Participants) | 36 | 65 | 0 | 0
  Week 12 | -17.44 (15.11) | -14.44 (13.96) |  |

6. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) at Week 12
Description: The DAS28 is a combined index for measuring disease activity in RA; the "28" refers to the number of joints included in the assessment. The index includes swollen and tender joint counts, acute phase response, and general arthritis disease activity status. An overall disease activity score of 5.1 or greater implies active disease, less than 3.2 implies low disease activity, and less that 2.6 implies disease remission.
Time Frame: Baseline, Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 72 | 9 | 97
Units on a scale
  Baseline: number analyzed (Participants) | 37 | 69 | 9 | 97
  Baseline | 6.29 (0.78) | 6.28 (1.03) | 5.42 (1.63) | 5.82 (1.28)
  Week 12: number analyzed (Participants) | 37 | 65 | 0 | 0
  Week 12 | -1.62 (1.28) | -1.15 (1.06) |  |

7. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission at Week 12
Description: as for outcome 6
Time Frame: Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Number; unit: Percent
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 66 | 9 | 97
Percent | 0 | 1.4 | 0 | 0

8. Secondary Outcome: Percentage of Participants Achieving CDAI Remission at Week 12
Description: The CDAI for Rheumatoid Arthritis (RA) assesses the severity of the disease using clinical data. It consists of the Patient Global disease Activity (PGA) estimate and the Evaluator Global disease Activity (EGA) estimate, each of which represent assessments of disease activity on a scale of 1-10, with 10 being maximum activity. CDAI remission is defined as a score of less than or equal to 2.8.
Time Frame: Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Number; unit: Percent
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 66 | 9 | 97
Percent | 0 | 1.4 | 0 | 0

9. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 12
Description: The ACR20 is a composite measure defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP). The ACR is reported as percent improvement at discrete time points.
Time Frame: Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Number (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 72 | 9 | 97
Percent | 43.2 [29.55 to 57.94] | 27.8 [19.42 to 37.88] | 0 [0.00 to 30.89] | 11.3 [6.66 to 18.32]

10. Secondary Outcome: Percentage of Participants Achieving ACR70 Response at Week 12
Description: The ACR70 is a composite measure defined as both improvement of 70% in the number of tender and number of swollen joints, and a 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP). The ACR is reported as percent improvement at discrete time points.
Time Frame: Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Number (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 72 | 9 | 97
Percent | 0 [0.00 to 9.15] | 1.4 [0.10 to 7.04] | 0 [0.00 to 30.89] | 0 [0.00 to 3.65]

11. Secondary Outcome: Change From Baseline in Simple Disease Activity Index (SDAI) Score at Week 12
Description: The SDAI consists of 5 parameters used to assess RA disease activity: 28-joint count assessments of tenderness and swelling, participant and investigator global assessments, and CRP levels. A composite score is produced, with remission defined as an SDAI of <3.3, low disease activity as ≤11, moderate disease activity as ≤26 and high disease activity as >26.
Time Frame: Baseline, Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 72 | 9 | 97
Scores on a scale
  Baseline: number analyzed (Participants) | 37 | 69 | 9 | 97
  Baseline | 38.84 (10.58) | 39.02 (14.55) | 31.23 (15.25) | 34.08 (16.69)
  Week 12: number analyzed (Participants) | 34 | 65 | 9 | 97
  Week 12 | -17.48 (14.48) | -14.99 (15.19) | -15.33 (18.24) | -13.15 (14.56)

12. Secondary Outcome: Change From Baseline in the Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The HAQ-DI is a 20-item, validated questionnaire used to assess difficulty in performing activities of daily living. The questionnaire assesses eight domains of physical functioning: Dressing and Grooming (2 items), Hygiene (3 items), Arising (2 items), Reach (2 items), Eating (3 items), Grip (3 items), Walking (2 items), Common Daily Activities (3 items). The questions assess usual abilities ranging from 0 "without any difficulty" to 3 "unable to do." A lower HAQ-DI score indicates better quality of life. Subscale scores are combined and the mean value is reported for each arm per timepoint.
Time Frame: Baseline, Week 12 of PoC and Week 12 of Extension Period Analysis (overall study week 24)
Population: The efficacy population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 37 | 72 | 9 | 97
Units on a scale
  Baseline: number analyzed (Participants) | 37 | 70 | 9 | 96
  Baseline | 1.63 (0.64) | 1.61 (0.76) | 1.29 (0.70) | 1.59 (0.71)
  Week 12: number analyzed (Participants) | 37 | 65 | 6 | 81
  Week 12 | -0.15 (0.52) | -0.24 (0.51) | -0.21 (0.74) | -0.21 (0.49)

13. Secondary Outcome: Serum RO7123520 Concentration
Time Frame: Pre-dose (0 hour), 1 hour post infusion (duration of infusion: approximately 1 hour) on Days 1, 14, 28, 56; Pre-dose (0 hour) on Days 84, 112
Population: All enrolled participants were included in the PK population. No PK analysis was performed due to an insufficient number of available participant samples for processing.
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Synovial Fluid RO7123520 Concentration
Time Frame: Pre-dose (0 hour) on Days 1, 84
Population: as for outcome 13
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to last participant last visit (approximately 2 years)
Description: The safety population included participants who received at least one dose of study drug.
Arm/Group | Placebo | Proof of Concept: RO7123520 810mg/Dose | Extension Period Analysis: RO7123520 360mg/Dose | Extension Period Analysis: RO70123520 810mg/Dose
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/70 | 0/9 | 0/97
Serious Adverse Events (participants affected / at risk) | 1/37 | 1/70 | 1/9 | 0/97
Other Adverse Events (participants affected / at risk) | 10/37 | 10/70 | 6/9 | 17/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | Proof of Concept: RO7123520 810mg/Dose (N=70) | Extension Period Analysis: RO7123520 360mg/Dose (N=9) | Extension Period Analysis: RO70123520 810mg/Dose (N=97)
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | Proof of Concept: RO7123520 810mg/Dose (N=70) | Extension Period Analysis: RO7123520 360mg/Dose (N=9) | Extension Period Analysis: RO70123520 810mg/Dose (N=97)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 9
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 2 | 0 | 0 | 0
Computerised tomogram abnormal (Investigations) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was prematurely terminated due to a lack of efficacy of the investigational drug. There were no serious safety issues or adverse events contributing to the decision to terminate early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03001219/Prot_SAP_000.pdf